CLINICAL TRIAL: NCT05847023
Title: Linguistic Underpinnings of Narrative in Aphasia (LUNA): A Proof-of-concept Study of a Novel Discourse Treatment for Aphasia Using Personal Narratives
Brief Title: Proof-of-concept Study of LUNA Intervention in Aphasia
Acronym: LUNA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City, University of London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TSA2017/01
Record Dates: First submitted 2023-03-27; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Aphasia; Stroke
Keywords: Treatment; Feasibility study; Discourse
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Intervention Model Description: The study is a single-blind, waitlist, randomised controlled trial of LUNA for people with chronic post-stroke aphasia. Participants will complete assessments at three time points: T1 (weeks 1&2), T2 (weeks 13 & 14) and T3 (weeks 25 & 26). Following T1, participants will be randomised to an immediate or delayed condition. Those in the immediate condition will receive LUNA therapy between T1 and T2. Those in the delayed condition will receive LUNA therapy between T2 and T3. All participants will be invited to participate in in-depth individual semi-structured interviews post-therapy to explore their experiences of taking part in the study.
Who Masked: Outcomes Assessor
Masking Description: The LUNA Assessors (2 staff) were blinded to group allocation throughout the study. The statistician leading on analysis of initial efficacy findings was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate LUNA intervention (Experimental): LUNA intervention between T1 and T2. No treatment between T2 and T3. LUNA intervention comprises 20hrs of face-to-face treatment, 2 sessions per week of 60 minutes each, for 10 weeks. One session is delivered by a qualified speech and language therapist; the other session is delivered by an assistant (student or volunteer) following guidance and under distance supervision. Both therapist and assistant will receive LUNA training. The treatment is specified in the TIDIER checklist. In brief, it aims to improve spoken discourse production, using personal narratives as assessment and treatment stimulate, and by integrating word, sentence and discourse level tasks. Treatment is manualised and has been codesigned with key stakeholders (providers and users).
  Interventions: Behavioral: LUNA
- Delayed LUNA intervention (Experimental): Wait between T1 and T2. LUNA between T2 and T3. LUNA intervention as above
  Interventions: Behavioral: LUNA

INTERVENTIONS:
Behavioral: LUNA — see description above

SUMMARY:
Existing evidence-based treatments for word-level and sentence-level impairments following aphasia typically do not generalise to gains in everyday communication for people with aphasia (after stroke). Novel treatments need to be developed to address this. LUNA is a novel multi-level discourse treatment for people with mild to moderate aphasia that addresses personal narratives in a personalised and meta-linguistic and metacognitive manner. This is a feasibility randomised waitlist controlled trial of LUNA, in 28 people with post-stroke chronic aphasia. It will test feasibility, acceptability, preliminary efficacy, and treatment fidelity. Findings will enable the investigators to judge whether there is merit in proceeding to a larger definitive trial.

DETAILED DESCRIPTION:
One third of stroke survivors have aphasia (a language impairment) which negatively affects communication, relationships, work, socialising, and wellbeing. Speech and language therapy is effective at improving language outcomes for people with aphasia (PWA) but gains in saying words and sentences rarely translate into gains in everyday talking (discourse). Most evidence generated over the last 40 years does not consider how words, sentences and everyday talk are linked together. Recent research signals new approaches are needed targeting multiple levels of language within the same treatment, and treatment needs to explicitly target everyday talking. Research conducted with stakeholders confirms new discourse treatments are a priority to clinicians and researchers, and improved everyday talking is prioritised by PWA as an outcome from rehabilitation.

The proposed research addresses the gap in the evidence base for a theoretically-underpinned multilevel discourse treatment for PWA. The project is titled LUNA and stands for Linguistic Underpinnings of Narrative in Aphasia. It focusses on personal narratives, that is, the short stories people tell others e.g. about recent holiday, funniest memory from school/ work, memorable life moments, etc. Personal stories are central to everyday talking; are important in health, recovery and adjustment; and are commonly used in clinical practice i.e. 70% of speech and language therapists (SLTs) the investigators surveyed in the United Kingdom ask patients to tell personal stories during rehabilitation. LUNA draws on existing word and sentence level treatments that are known to be effective in improving language. The discourse literature is less developed, but describes strategies that similarly feature in LUNA treatment (e.g. telling the key elements of a story and doing so in the correct order so the listener understands). LUNA integrates these and works directly with the participant to improve their own stories. Choosing personalised vocabulary (i.e. the person's own words) increases motivation. Finally, LUNA teaches the person about their language, so they understand their difficulties, thereby empowering them to make connections from clinic to their real life use of talking.

In response to the COVID 19 crisis the investigators plan to conduct all data collection remotely, via video conferencing technology. There is growing evidence that telehealth can be employed successfully in aphasia rehabilitation. Remote administration of aphasia assessment has been shown to be valid, reliable and acceptable to people with aphasia. While not extensively tested, remote therapy has also proved feasible and has produced outcomes that are similar to those achieved by face to face delivery. This study aims to add to the evidence for aphasia tele-rehabilitation by testing the first application of remote discourse therapy.

Aims:

This study will test feasibility of LUNA in terms of participant recruitment and retention, and adherence throughout the study (assessment and treatment sessions). It will explore participant acceptability of LUNA and project procedures (satisfaction, perceived benefits, assessment and treatment burden) in semi-structured individual interviews with participants.

It will investigate initial efficacy by comparing outcomes on a range of measures across participants who have and have not received LUNA intervention. It will assess treatment fidelity by reviewing a sample of videotaped sessions to check they were delivered as intended by the treatment manual. The study will also test the feasibility and acceptability of remote assessment and treatment delivery. For example, recruitment, retention and compliance data will attempt to identify losses due to technological factors; and interview questions will explicitly probe the experience of using video-conferencing technology.

Indicative outcome data will be for remote (not face-to-face) LUNA.

Design:

The study is a single-blind, waitlist, randomised controlled trial of LUNA for people with chronic post-stroke aphasia. Participants will complete assessments at three time points: T1 (weeks 1&2), T2 (weeks 13 & 14) and T3 (weeks 25 & 26). Following T1, participants will be randomised to an immediate or delayed condition. Those in the immediate condition will receive LUNA therapy between T1 and T2. Those in the delayed condition will receive LUNA therapy between T2 and T3. All participants will be invited to participate in in-depth individual semi-structured interviews post-therapy to explore their experiences of taking part in the study.

In line with selection criteria, participants will not be receiving any other speech and language therapy during the study. Owing to COVID 19, it is anticipated that most participants will not have access to usual care (attendance at stroke groups). Some may access on-line supports, for example provided by Aphasia Re-Connect. Use of such services is not an exclusion criterion. Use of other services will be explored in the interviews.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of ischaemic or haemorrhagic stroke
* have aphasia due to a stroke that occurred at least 12 months prior to recruitment
* literate and fluent users of English prior to their stroke (self-reported)
* have adequate hearing and vision with aids and glasses, e.g. in order to see pictorial and written assessment and therapy materials
* must have access to a computer or tablet and an internet connection
* must be able to download and access Zoom, either independently or with the support of a friend/family member who is living with them

Exclusion Criteria:

* must not be receiving speech and language therapy elsewhere for the duration of the study. Usual stroke supports, for example provided by the voluntary sector, can proceed, although these are likely to be curtailed owing to COVID-19
* must not be participating in any other aphasia treatment research project for the duration of the study
* must not have severe aphasia, defined as a score of 7 or less on the Frenchay Aphasia Screening Test (FAST: Enderby et al., 1986; unlikely to benefit from treatment)
* must not have a secondary cognitive diagnosis such as dementia. This will be established via self-report and the confirmation of the group co-ordinator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Personal narratives measure (LUNA Discourse Protocol) | Change from baseline (T1: weeks 1 and 2) to immediately post treatment (T2: weeks 13 and 14) to follow up (T3: weeks 25 and 26)
  Participants will produce two personal narratives at each assessment point, which will be video/audio recorded. They will be given instructions e.g. length of narrative, indication of topic etc. The narrative will be spoken face-to-face to the assessing therapist. S/he will not provide any cues or ask questions. Recording will cease when the participant indicates that the story is finished. Discourse samples will be analysed according to the LUNA Research Discourse Analysis Protocol. The analysis yields the following data: number and %narrative words, and number of narrative words/minute; %Correct Information Units( CIU); number of CIUs/minute; %complete utterances; %single versus multi-clause utterances; #1, 2, and 3 argument utterances; Predicate Argument Score; story grammar count of elements; global coherence score; local coherence score; reference chains count; and overall listener judgment. Number of narrative words is proposed as the primary discourse outcome.

SECONDARY OUTCOMES:
The Western Aphasia Battery-Revised Aphasia Quotient (WAB-R AQ) | Change from baseline (T1: weeks 1 and 2) to immediately post treatment (T2: weeks 13 and 14) to follow up (T3: weeks 25 and 26)
  Tests speaking, auditory comprehension, naming and repetition across 4 sections. Takes 30-45 minutes. Internationally used language functioning test; also recommended internally as a core outcome measure. Provides information on type of aphasia, and severity.
The Communicative Participation Item Bank (CPIB) - General Short Form [Patient Reported Outcome Measure] | Change from baseline (T1: weeks 1 and 2) to immediately post treatment (T2: weeks 13 and 14) to follow up (T3: weeks 25 and 26)
  10 items. Items are worded as the degree to which the person's condition interferes with e.g. communicating when out in the community. Designed for adults with communication disorders with substantial input from individuals themselves. Short form recently proven appropriate for people with aphasia (Baylor et al., 2017). We anticipate overlap in item content of the CPIB with the ALA, however, we are intentionally including this instrument as it is possible that this much shorter instrument may be more acceptable (for its brevity) and on post-hoc analysis from the interviews, may align more with participants' perceptions of benefit from the intervention. This will contribute to decision-making for a future large trial. <15 minutes.
The Communication Confidence Rating Scale for Aphasia (CCRSA) [Patient Reported Outcome Measure] | Change from baseline (T1: weeks 1 and 2) to immediately post treatment (T2: weeks 13 and 14) to follow up (T3: weeks 25 and 26)
  10 items. The only confidence measure in our field. Increasingly used in treatment studies. Takes <10minutes.
The Assessment for Living with Aphasia (ALA) [Patient Reported Outcome Measure] | Change from baseline (T1: weeks 1 and 2) to immediately post treatment (T2: weeks 13 and 14) to follow up (T3: weeks 25 and 26)
  52 items. Is a pictographic self-report test of aphasia-related quality of life. Created by internationally leading charity in Canada. Increasingly used in treatment studies. Takes up to 45 minutes.
Visual Analogue Mood Scales (VAMS) [Patient Reported Outcome Measure] | Change from baseline (T1: weeks 1 and 2) to immediately post treatment (T2: weeks 13 and 14) to follow up (T3: weeks 25 and 26)
  Following feedback from our advisors with aphasia (and supported by the research team), a single item mood measure, the Visual Analogue Mood Scales (VAMS) Sad scale (Stern et al., 1997) was added to all testing time points. It has been used successfully in aphasia studies (Marshall et al., 2019; Thomas et al., 2013) and takes 3 minutes to complete. It is accessible and appropriate to be used with stroke survivors who have aphasia. Content validity has been established (Nyenhuis et al., 1997; Stern et al., 1997) and test re-test reliability (House et al., 2012).

OTHER OUTCOMES:
Percentage of those eligible who consent | Week 27
  Feasibility of recruitment was calculated by the number of the participants who consented, divided by the number those who met eligibility criteria, multiplied by 100.
Percentage of retention | Week 27
  Feasibility of retention to the trial was calculated by the number of participants available at follow up (week 25 and 26), divided by the total consented, multiplied by 100.
Percentage of treatment sessions attended with reasons for non-attendance | Week 27
  Acceptability of the intervention to participants was calculated by the number of treatment sessions attended as planned (at the time and date arranged), divided by total treatment sessions offered, multiplied by 100.
Rates of missing data | Week 27
  Acceptability of outcome measures was calculated by the number of missing data points.
Presence of floor or ceiling effects | Week 27
  Appropriateness of outcome measures was also informed by the presence of floor or ceiling effects, defined as more than 15% of participants scoring the lowest or highest score.
Estimating sample size | Week 27
  Means, standard deviations and effect sizes of the proposed primary clinical outcome measures and retention rates
Assessing treatment fidelity | Week 27
  Adherence to treatment manual was calculated for each checklist item as a percentage of present items.
In-depth qualitative interviews | Weeks 25 and 26
  Interview data will illuminate participants' views about the intervention, the study experience and procedures.
The Session Rating Scale | Weeks 25 and 26
  A four item rating scale of therapeutic alliance. It asks participants to rate if they felt listened to, if the therapy was important, if they liked it and the overall fit. Scores range from 0-10 where 10 represents high therapeutic alliance. The scale has demonstrated high internal consistency and moderate test-retest reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Cruice, Principal Investigator — City, University of London; Prof Dipper, Principal Investigator — City, University of London
Locations (1):
- Department of Language and Communication Science, City, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agostini M, Garzon M, Benavides-Varela S, De Pellegrin S, Bencini G, Rossi G, Rosadoni S, Mancuso M, Turolla A, Meneghello F, Tonin P. Telerehabilitation in poststroke anomia. Biomed Res Int. 2014;2014:706909. doi: 10.1155/2014/706909. Epub 2014 Apr 15. PMID 24829914
- [Background] Brady MC, Kelly H, Godwin J, Enderby P. Speech and language therapy for aphasia following stroke. Cochrane Database Syst Rev. 2012 May 16;(5):CD000425. doi: 10.1002/14651858.CD000425.pub3. PMID 22592672
- [Background] Cruice, M., Woolf, C., Caute, A., Monnelly, K., Wilson, S. & Marshall, J. (2021) Preliminary outcomes from a pilot study of personalised online supported conversation for participation intervention for people with Aphasia, Aphasiology, 35:10, 1293-1317, DOI: 10.1080/02687038.2020.1795076
- [Background] Dekhtyar M, Braun EJ, Billot A, Foo L, Kiran S. Videoconference Administration of the Western Aphasia Battery-Revised: Feasibility and Validity. Am J Speech Lang Pathol. 2020 May 8;29(2):673-687. doi: 10.1044/2019_AJSLP-19-00023. Epub 2020 Mar 19. PMID 32191122
- [Background] Enderby P, Wood V, Wade D. Frenchay aphasia screening test (FAST). West Sussex: Wiley; 1986.
- [Background] Guo YE, Togher L, Power E, Hutomo E, Yang YF, Tay A, Yen SC, Koh GC. Assessment of Aphasia Across the International Classification of Functioning, Disability and Health Using an iPad-Based Application. Telemed J E Health. 2017 Apr;23(4):313-326. doi: 10.1089/tmj.2016.0072. Epub 2016 Nov 1. PMID 27802112
- [Background] Julious, S.A. (2005), Sample size of 12 per group rule of thumb for a pilot study. Pharmaceut. Statist., 4: 287-291. https://doi.org/10.1002/pst.185
- [Background] Rose M, Ferguson A, Power E, Togher L, Worrall L. Aphasia rehabilitation in Australia: Current practices, challenges and future directions. Int J Speech Lang Pathol. 2014 Apr;16(2):169-80. doi: 10.3109/17549507.2013.794474. Epub 2013 Jun 18. PMID 23777446
- [Background] Theodoros D, Hill A, Russell T, Ward E, Wootton R. Assessing acquired language disorders in adults via the Internet. Telemed J E Health. 2008 Aug;14(6):552-9. doi: 10.1089/tmj.2007.0091. PMID 18729754
- [Background] Wallace SJ, Worrall L, Rose T, Le Dorze G, Cruice M, Isaksen J, Kong APH, Simmons-Mackie N, Scarinci N, Gauvreau CA. Which outcomes are most important to people with aphasia and their families? an international nominal group technique study framed within the ICF. Disabil Rehabil. 2017 Jul;39(14):1364-1379. doi: 10.1080/09638288.2016.1194899. Epub 2016 Jun 27. PMID 27345867
- [Background] J. Webster, A. Whitworth & J. Morris (2015) Is it time to stop "fishing"? A review of generalisation following aphasia intervention, Aphasiology, 29:11, 1240-1264, DOI: 10.1080/02687038.2015.1027169
- [Background] Weidner, K., & Lowman, J. (2020). Telepractice for adult speech-language pathology services: A systematic review. Perspectives of the ASHA Special Interest Groups, 5(1), 326-338. doi:10.1044/2019_PERSP-19-00146
- [Background] A. Whitworth, S. Leitão, J. Cartwright, J. Webster, G.J. Hankey, J. Zach, D. Howard & V. Wolz (2015) NARNIA: a new twist to an old tale. A pilot RCT to evaluate a multilevel approach to improving discourse in aphasia, Aphasiology, 29:11, 1345-1382, DOI: 10.1080/02687038.2015.1081143
- [Background] Woolf C, Caute A, Haigh Z, Galliers J, Wilson S, Kessie A, Hirani S, Hegarty B, Marshall J. A comparison of remote therapy, face to face therapy and an attention control intervention for people with aphasia: a quasi-randomised controlled feasibility study. Clin Rehabil. 2016 Apr;30(4):359-73. doi: 10.1177/0269215515582074. Epub 2015 Apr 24. PMID 25911523
- [Background] Cruice M, Botting N, Marshall J, Boyle M, Hersh D, Pritchard M, Dipper L. UK speech and language therapists' views and reported practices of discourse analysis in aphasia rehabilitation. Int J Lang Commun Disord. 2020 May;55(3):417-442. doi: 10.1111/1460-6984.12528. Epub 2020 Feb 24. PMID 32090417
- [Background] Dipper, L., Marshall, J., Boyle, M., Botting, N., Hersh, D., Pritchard, M., & Cruice, M. (2021) Treatment for improving discourse in aphasia: a systematic review and synthesis of the evidence base, Aphasiology, 35:9, 1125-1167, DOI: 10.1080/02687038.2020.1765305
- [Derived] Dipper L, Devane N, Barnard R, Botting N, Boyle M, Cockayne L, Hersh D, Magdalani C, Marshall J, Swinburn K, Cruice M. A feasibility randomised waitlist-controlled trial of a personalised multi-level language treatment for people with aphasia: The remote LUNA study. PLoS One. 2024 Jun 14;19(6):e0304385. doi: 10.1371/journal.pone.0304385. eCollection 2024. PMID 38875279